CLINICAL TRIAL: NCT07352592
Title: Process-Based Approach Case Series For Anxiety Problems
Acronym: PBT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nicholas C. Borgogna, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300016048
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Anxiety
Keywords: PBT; PBA; Process-Based Approach; Process-Based Cognitive Behavioral Therapy; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Process-based approach (Experimental): PBA therapy
  Interventions: Behavioral: Process-Based Approach

INTERVENTIONS:
Behavioral: Process-Based Approach — Process-Based Approaches (PBA) were developed to improve psychotherapy outcomes. Early writings referred to PBA as process-based therapy or process-based cognitive behavioral therapy. The current nomenclature was adopted to distinguish PBA as a unifying approach that incrementally builds on clinical psychological science rather than a manualized treatment protocol. PBA provides a framework for flexibly applying evidence-based techniques from multiple therapeutic traditions to target hypothesized psychological processes that give rise to individual patient presentations. Each patient is conceptualized independently, and intervention structure may vary substantially based on need, while retaining empirically supported tools. This contrasts with disorder-specific treatment manuals, which assume homogeneity despite substantial variability in underlying processes (e.g., anxiety).
  Other Names: PBT

SUMMARY:
A case series of PBA intervention for anxiety problems.

DETAILED DESCRIPTION:
Participants will self-refer to this study by emailing a research assistant (Mr. Whittington).

They will then attend a screening session where they complete an informed consent form and are assessed for inclusion/exclusion criteria. During the screening the research assistant will conduct a clinical interview and collaboratively identify hypothetical processes (e.g. avoidance) that might be contributing to the participants anxiety symptoms. Together, they will identify 8-items from the process-based assessment tool (see survey) that might be relevant to the participants anxiety.

Participants will then complete a baseline survey battery on a lab computer (via Qualtrics; ~20 minutes).

Participants will then complete a two-week assessment period where they complete brief (<2 minute) surveys five times a day (approximately 9 am, noon, 2 pm, 5 pm, and 8 pm) each day for the two weeks. These surveys will be sent to participants' phone via Qualtrics. These surveys will be the 8-items identified during the intake session, with one additional item assessing momentary anxiety and an additional item assessed momentary quality of life perception.

The research team will use the data gathered during the two-week assessment period to create personalized networks of processes leading to participant anxiety symptoms. Each participants' network will guide their therapy treatment.

Participants will then attend up to 25 sessions of counseling for their anxiety. Sessions will occur roughly weekly and will last approximately 50 minutes. All sessions will occur in Dr. Borgogna's lab and clinic space (Campbell Hall Ste 310) on the UAB campus. The therapists in the study will all be masters-level clinicians in the UAB medical/clinical psychology program preparing for licensure (Mr. Whittington, Mr. Johnson, and Ms. Jafari) or a licensed clinical psychologist (Dr. Borgogna). Therapy sessions for pre-licensed clinicians will be recorded onto a UAB computer in Dr. Borgogna's lab and reviewed for supervision purposes by Dr. Borgogna (A/V recordings not for research purposes). Recordings will be deleted within 30 days of each therapy session.

Participants will complete the main battery again at post-test.

ELIGIBILITY:
Inclusion Criteria:

* Score on GAD-7 >10 at baseline
* Access to mobile device

Exclusion Criteria:

* Current psychotherapy treatment
* Current/past severe psychopathology (e.g., history of psychosis, suicide attempt or self-injury within the past 12 months, narcotics use within the past 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder-7 | From enrollment to the end of treatment, up to 25 weeks.
  Anxiety scale
Beck Anxiety Inventory | From enrollment to the end of treatment, up to 25 weeks.
  Anxiety Measure

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | From enrollment to the end of treatment, up to 25 weeks.
  Depression measure
Experiential Avoidance Rating Scale | From enrollment to the end of treatment, up to 25 weeks.
  Experiential avoidance measure
Quality of Life Scale | From enrollment to the end of treatment, up to 25 weeks.
  Quality of Life Measure
Big Five Inventory | From enrollment to the end of treatment, up to 25 weeks.
  Measure of Personality
PSY-Flex | From enrollment to the end of treatment, up to 25 weeks.
  Psychological flexibility measure

OTHER OUTCOMES:
Process-based assessment tool | Five times a day for two weeks prior to intervention
  A collection of hypothetical processes that might be correlated with mental illness outcomes. Selections will be used to inform patient conceptualizations prior to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Borgogna, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: Yes
De-identified outcome scores will be shared in publication. Raw scores are available upon request to the principal investigator.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 2027-2030
Access Criteria: PhD-level researchers associated with academic institutions will have access to de-identified spreadsheets and code.